CLINICAL TRIAL: NCT04846010
Title: Treating Sequalae Caused by Post-acute Sequelae of SARS (Severe Acute Respiratory Syndrome)-CoV-2 Infection
Brief Title: Recovering Damaged Cells for Sequelae Caused by COVID-19, SARS-CoV-2
Acronym: sequelae
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All Natural Medicine Clinic, LLC (Other)
Responsible Party: Principal Investigator, Wanzhu Hou, President, All Natural Medicine Clinic, LLC
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHM2282395-2
Record Dates: First submitted 2021-03-31; First posted 2021-04-15 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Sequelae of; Infection; Post Infection Glomerulonephritis; Post-Infectious Peripheral Neuralgia; Post-Infectious Disorder (Disorder); Post-Infectious Arthritis; Post-Infectious Polyneuritis; Post-Infectious Parkinsonism; Post-Infectious Hypothyroidism; Post Infectious Osteoarthritis; Anxiety Disorders; Depression; Depression, Anxiety; Depression, Bipolar; Insomnia; GERD; Gastro Esophageal Reflux; Hepatitis; Glomerulonephritis
Keywords: treatment of Covid-19 virus infection; COVID stress syndrome; COVID19 stress syndrome; sequelae; sequels; loss of smell; loss of taste; emotion disorder; panic disorder; Post-Traumatic Stress Disorder (PTSD); Depression; Anxiety; Heartburn; GERD; Gastroesophageal reflux disease; Sleep Disorders
MeSH Terms: conditions — Infections; Post-Infectious Disorders; Arthritis, Reactive; Guillain-Barre Syndrome; Anxiety Disorders; Depression; Bipolar Disorder; Sleep Initiation and Maintenance Disorders; Gastroesophageal Reflux; Hepatitis; Glomerulonephritis; COVID-19 stress syndrome; Anosmia; Ageusia; Panic Disorder; Stress Disorders, Post-Traumatic; Heartburn; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: This clinical study designed with a sequential assignment: participants receive their medical herbs depending on their pathological states; through one course of the treatment, we will review their symptoms and corresponding indicators of visceral damage。
Masking Description: To restore the damaged structure and function of cells, participants come for the treatment with their diagnosis and experiment medics from their conventional practitioners. There have no masking for anybody.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- antigen (Active Comparator): The antigen is the cell that is destroyed by inflammation, which can perform as swollen, fatty, apoptosis, necrosis, and lethal pathological states. Some pathological cells can be saved and returned to customary conditions, like swollen, fatty, early apoptosis, but necrosis, lethal.
  Interventions: Combination Product: PurWet; Combination Product: FurFat; Combination Product: PurApo; Combination Product: PurPhl
- Internal environment (Active Comparator): The internal environment is critical to the damaged cells recovering. Mainly it is covered by two major parts: metabolites and thrombus.
  Interventions: Combination Product: PurClo
- Communication between cells (Active Comparator): The communication between organs, cells, helps the damaged cells recover and reduce symptoms.
  Interventions: Combination Product: PurInf; Combination Product: Smoliv

INTERVENTIONS:
Combination Product: PurWet — (1) cang zhu (Atractylodis Rhizoma), bai (zhu Atractylodis macrocephalae Rhizoma), dang shen (Codonopsis Radix), huang qi (Astragali Radix), Fu ling (Poria), Zhu ling (polyporus), Ze xie (Alismatis Rhizoma), Yi yi ren (Coicis Semen), gan cao (Glycyrrhizae Radix),
  Arms: antigen
Combination Product: FurFat — (2).shan zha (Crataegi Fructus), Jue Ming Zi (Cassiae Semen), He ye (Nelumbinis Folium), Da huang (Rhei Radix et Rhizoma), Ze xie (Alismatis Rhizoma), dan shen ( Salviae miltiorrhizae Radix).
  Arms: antigen
Combination Product: PurApo — (3)Sheng Di Huang (Rehmanniae Radix), Xuan Shen (Scrophulariae Radix), mai men dong (Ophiopogonis Radix), shan zhu yu (Corni Fructus), shan yao (Dioscoreae Rhizoma), sha yuan zi (Astragali complanati Semen), ci ji li (Tribuli Fructus), nu zhen zi (Ligustri lucidi Fructus)
  Arms: antigen
Combination Product: PurPhl — (4) chen pi (Citri reticulatae Pericarpium), hua ju hong (Citri grandis Exocartium rubrum), zhi shi (Aurantii Fructus immaturu), zhi ban xia (Pinelliae Rhizoma preparatum), zhi tian nan xing (Arisaematis Rhizoma preparatum),sha ren (Amoni Fructus), Gua lou (Trichosanthis Fructus), Chuan bei mu ( Fritillatiae cirrhosae Bulbu), Fu ling ( Poria), Da huang ( Rhei Radix et Rhizoma).
  Arms: antigen
Combination Product: PurClo — (2) Dan shen (Salviae miltiorrhizae Radix), Yu jin (Curcumae Radix), chi shao (Paeoniae Radix rubra), tao ren (Persicae Semen), hong hua (Carthami Flos)
  Arms: Internal environment
Combination Product: PurInf — (1) lei gong teng (Tripterygii wilfordii Radix), Huang Qin (Scutellariae Radix), Huang Lian (Coptidis Rhizoma), Huang Bai (Phellodendri Cortex), Zhi Zi (Gardeniae Fructus).
  Arms: Communication between cells
Combination Product: Smoliv — (2). Vagus never communicates with LES: yu jin (Curcumae Radix), Chai Hu (Bupleuri Radix), chi shao (Paeoniae Radix rubra), Mu Dan Pi (Moutan Cortex), chuan lian zi (Toosendan Fructus), long gu (Fossilia Ossis Mastodi), mu li (Ostreae Concha)
  Arms: Communication between cells

SUMMARY:
Post-acute sequelae of SARS-CoV-2 infection can cause multiple system function disorders, and complicated symptoms last for an extended period. The virus can cause this continued infection, or the virus causes immune system function disorder and post-infectious autoimmune disease. The clinical symptoms can be smell loss, taste loss to liver function disorder, kidney function failure, different. No matter how complicated the systems showed in the clinic, all of the symptoms are due to the specific cells being damaged. Our clinical study is focused on recovering the damaged structure and function of the cells that could restore the organ function back to normal or close to normal

DETAILED DESCRIPTION:
SARS-CoV-2 caused sequela is a pathological condition, and specific cells are damaged from a prior disease, injury, or attack. Post-Acute Sequelae of SARS-CoV-2 Infection (PASC) is caused by an infection of SARS-CoV-2 and COVID-19 virus. The virus or virus-triggered disorder immunity attacks target tissue(s) and organ(s). No matter name of the virus and the cells, tissue(s), or organ(s), they all belong to the category of antigen and cause an immune response; this can induce inflammation or not depending on the immune system tolerance . While older patients may have an increased risk of developing severe disease or sequelae, young survivors have also reported symptoms months after acute infection of SARS-CoV-2, reported by the British Lung Foundation. Some infected people, referred to as long-haulers, experience a long period of symptoms. Characterization of the etiology and pathophysiology of late sequelae is underway and may reflect organ damage from the acute infection phase; manifestations of a persistent hyperinflammatory state even perform as autoimmune diseases. Rheumatic disease can also occur during the infection of COVID. Ongoing viral activity indicates an inadequate antibody response. Factors in addition to acute illness that may further complicate the picture include physical deconditioning at baseline or after a long disease course, pre-COVID-19 comorbidities, and psychological sequelae following a long or difficult disease course relating to lifestyle changes due to the pandemic. Likely, the persistent sequelae of COVID-19 represent multiple syndromes resulting from distinct pathophysiological processes along the spectrum of disease. So far, no specific medicine has been identified for treating the COVID-19 virus and post-acute sequelae of SARS-CoV-2. Due to the difficulty treating either SARS-CoV-2 or its caused sequelae, there is a very pessimistic suggestion: People must live with COVID-19 forever. Most people who contract coronavirus disease 2019 (COVID-19) infection recover entirely within a few weeks. However, the long-haulers continue to experience symptoms after their initial recovery. This condition has been called post-COVID-19 syndrome or "long COVID-19." Older people and people with many severe medical conditions are the most likely to experience lingering COVID-19 symptoms, but even young, otherwise healthy people can feel unwell for weeks to months after infection. The most common signs and symptoms that linger over time include fatigue, shortness of breath, cough, joint pain, and chest pain. Other long-term signs and symptoms may include muscle pain or headache, fast or pounding heartbeat, loss of smell or taste, memory and concentration or sleep problems, and rash or hair loss, the Mayo Clinic reported.

Virus infections have been long associated with autoimmune diseases, whether multiple sclerosis, diabetes, or myocarditis. Three potential mechanisms for virus-induced autoimmune disease or virus-induced immunopathology are molecular mimicry, bystander activation, and persistent virus infection.

Those prolonged symptoms are consistent with the internal physical pathological process. That can be the virus infection continuing, or the infection triggered an immune reaction in one or more physical locations when a person became infected with the COVID-19 virus.

Here is the critical point: when the structure of cells is destroyed, the result is the affected cell's function will be lost. Does the etiology directly destroy the antigen, or the virus trigger the disorder immunity to destroy the antigen? The results are the same: the antigen is under inflammation. Returning the damaged cells (antigen) to normal or close to normal states is the key to saving lives.

This raises questions concerning how can we protect those cells from becoming damaged and how can we return injured cells to their normal function? Regardless of whether the cell has been damaged directly by the virus infection, or another reason like disordered immunity, my clinical research will show how to solve those medical problems.

ELIGIBILITY:
Inclusion Criteria:

* The participants must receive medical herbs as a treatment method;
* Participants are not limited by age, sex, race, or location;
* Participants are including infants;
* Participants are including pregnant woman;
* The participants had an infection history of SARS-CoV-2 in past one month;
* The participants provide SARS-CoV-s diagnoses (Molecular or Antigen). Test was *positive, now hold negative reports
* Participants hold reports of immune system medics, like immunoglobulin M (IgM), immunoglobulin G (IgG);
* Reports that is evidence of specific organ damaged, including assay reports or image reports
* Participants must agree to take medical herbs for at least 3 months as one course continually;
* Participants must agree to repeat the assay and image test to monitor the treatment results;
* Participants must report their Manifestations clearly to investigators;
* Participants must agree to continue the next course of the treatment after the evaluation if it is necessary;
* The treatment goal is to become symptom-free, and experiment assays went to normal

Exclusion Criteria:

* Participants don't want to take medical herbs;
* Participants have symptoms of sequelae but is not caused by SARS-CoV-2 (COVID-19);
* Participants have not symptoms after COVID-19 infection, no assays abnormal either;
* Participants don't want to repeat the experiment assays;
* Participants are in E.R. or ICU during the application or enrollment;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Monitoring symptoms | 3 months as a course
  Measuring the symptoms of chest pain, cough, loss of smell, loss of taste by Visual Analog Score (VAS)

SECONDARY OUTCOMES:
Monitoring emotion changing | 3 months as a course.
  measuring anxiety, depression, bipolar feeling by Visual Analog Score (VAS)
Checking heart burn symptom | 3 months as a course.
  Measuring stomach reflux symptom by Visual Analog Score (VAS)
Monitoring thyroid function | 3 months as a course
  Measuring thyroid hormone3, 4 (T3,T4), thyroid-stimulating hormone (TSH) level
Monitoring liver function | 3 months as a course
  Measuring alanine transaminase (ALT), Aspartate transaminase (AST), alkaline phosphatase (ALP) recovering
Monitoring kidney function | 3 months as a course
  Measuring estimated glomerular filtration rate (eGFR), creatinine (Cr.) level

CONTACTS AND LOCATIONS:
Overall Officials: Wanzhu Hou, CMD, Principal Investigator — All Natural Medicine Clinic, LLC
Locations (1):
- All Natural Medicine Clinic, LLC, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Medical herbs are not directing immunity only, but also recover the damaged structure and function of cells that be destroyed by inflammation. We will publish the process of the treatment as soon as we can.
Supporting Information: CSR
Time Frame: We will continually publish clinical case study online.
Access Criteria: If you are a conventional medical practitioner, you can open it, and you will experience the different practice in clinic.
  If you are a helictical medical practitioner, you can learn how integrative medicine practice in clinic.
URL: https://anmedicine.com/blog/

REFERENCES:
- [Background] Wanzhu Hou, et al. Treating Autoimmune disease with Chinses Medicine, Elsevier, 2011
- [Background] Wannzhu Hou Cellular Structure and its Function is the key for keeling Diseases, Certification and Registration number: TXu 1-938-144 July 30, 2014
- [Background] Zigmond E, Varol C, Farache J, Elmaliah E, Satpathy AT, Friedlander G, Mack M, Shpigel N, Boneca IG, Murphy KM, Shakhar G, Halpern Z, Jung S. Ly6C hi monocytes in the inflamed colon give rise to proinflammatory effector cells and migratory antigen-presenting cells. Immunity. 2012 Dec 14;37(6):1076-90. doi: 10.1016/j.immuni.2012.08.026. Epub 2012 Dec 6. PMID 23219392
- [Background] Jurewicz MM, Stern LJ. Class II MHC antigen processing in immune tolerance and inflammation. Immunogenetics. 2019 Mar;71(3):171-187. doi: 10.1007/s00251-018-1095-x. Epub 2018 Nov 12. PMID 30421030
- [Background] Wang F, Kream RM, Stefano GB. Long-Term Respiratory and Neurological Sequelae of COVID-19. Med Sci Monit. 2020 Nov 1;26:e928996. doi: 10.12659/MSM.928996. PMID 33177481
- [Background] Pollard CA, Morran MP, Nestor-Kalinoski AL. The COVID-19 pandemic: a global health crisis. Physiol Genomics. 2020 Nov 1;52(11):549-557. doi: 10.1152/physiolgenomics.00089.2020. Epub 2020 Sep 29. PMID 32991251
- [Background] Schvartz A, Belot A, Kone-Paut I. Pediatric Inflammatory Multisystem Syndrome and Rheumatic Diseases During SARS-CoV-2 Pandemic. Front Pediatr. 2020 Dec 4;8:605807. doi: 10.3389/fped.2020.605807. eCollection 2020. PMID 33344389
- [Background] Smatti MK, Cyprian FS, Nasrallah GK, Al Thani AA, Almishal RO, Yassine HM. Viruses and Autoimmunity: A Review on the Potential Interaction and Molecular Mechanisms. Viruses. 2019 Aug 19;11(8):762. doi: 10.3390/v11080762. PMID 31430946
- [Background] Ploumpidis D. Living with covid-19. Psychiatriki. 2020 Jul-Sep;31(3):197-200. doi: 10.22365/jpsych.2020.313.197. English, Greek, Modern. PMID 33099460
- [Background] Fujinami RS, von Herrath MG, Christen U, Whitton JL. Molecular mimicry, bystander activation, or viral persistence: infections and autoimmune disease. Clin Microbiol Rev. 2006 Jan;19(1):80-94. doi: 10.1128/CMR.19.1.80-94.2006. PMID 16418524
- [Background] Honda T, Egen JG, Lammermann T, Kastenmuller W, Torabi-Parizi P, Germain RN. Tuning of antigen sensitivity by T cell receptor-dependent negative feedback controls T cell effector function in inflamed tissues. Immunity. 2014 Feb 20;40(2):235-247. doi: 10.1016/j.immuni.2013.11.017. Epub 2014 Jan 16. PMID 24440150
- See also: Every disease happened on cell's level, recovering the damaged structure and function is the key for healing the sequelae that caused by COVID-19 virus infection — http://www.anmedicine.com